CLINICAL TRIAL: NCT06751472
Title: Long-Term Follow-up of the Effect of Conventional Radiofrequency Thermocoagulation Application to the Articular Branches of the Femoral and Obturator Nerve on Pain and Functional Capacity in Patients With Chronic Hip Pain
Brief Title: Long-Term Follow-up of Radiofrequency to Articular Branches of the Femoral and Obturator Nerve in Chronic Hip Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, Aydin Adnan Menderes University, Aydin Adnan Menderes University
Other Study IDs: 2024-218
Record Dates: First submitted 2024-12-23; First posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Conventional Radiofrequency Thermocoagulation Application to the Articular Branches of the Femoral and Obturator Nerve; Chronic Hip Pain
Keywords: chronic hip pain; radiofrequency thermocoagulation; Articular Branches of the Femoral and Obturator Nerve

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- RFT: Conventional radiofrequency thermocoagulation (RFT) procedure was applied to the femoral and obturator nerve joint branches electively due to chronic hip pain.
  Interventions: Diagnostic Test: VPS (Verbal Pain Score); Diagnostic Test: WOMAC (Western Ontario and McMaster Universities Arthritis Index) scale

INTERVENTIONS:
Diagnostic Test: VPS (Verbal Pain Score) — İt is a pain intensity determination system based on the system where there person tells a point between 0=(no pain) 10=( unbearable pain) and to describe their pain
Diagnostic Test: WOMAC (Western Ontario and McMaster Universities Arthritis Index) scale — It includes 24 questions under three sub-headings as pain, stiffness and physical function

SUMMARY:
It has been observed that the deterioration in the physical performance of the hip, the medical need before the specialist consultation and the deterioration in the health status can progress treatment[3]. When conservative treatment methods such as physical therapy and weight change, the use of walking aids (such as a cane) and analgesic agents are used, these interruptions usually provide short-term and partial benefits. After the application of medical treatment procedures, hip prostheses are usually separated. However, the additional diseases of the patients, the fact that the surgery is a major surgery and the mortality rate is high, and the life of the prostheses used are limited have led to the search for alternative pain palliation.

Hip joint radiofrequency thermocoagulation is a procedure performed in our clinic. In this study, we aimed to examine the long-term effects of hip RFT on pain and functional capacity changes in patients.

DETAILED DESCRIPTION:
After obtaining hospital ethics committee approval, it was planned to retrospectively examine adult patients over the age of 18 who applied to the outpatient clinic of the Department of Algology, ADÜTF, between May 2021 and September 2023 and who underwent elective conventional radiofrequency thermocoagulation (RFT) procedure to the articular branches of the femoral and obturator nerves due to chronic hip pain. The prospective studies conducted in our clinic titled "Treatment of chronic hip pain with conventional radiofrequency thermocoagulation to the articular branches of the femoral and obturator nerve" and "Comparison of Conventional Radiofrequency Thermocoagulation to the Articular Branches of the Femoral and Obturator Nerve in Chronic Hip Pain with Intra-Articular Steroid Injection and Pericapsular Nerve Group (PENG) Block" (theses of assistants Sevilay Şimşek Karaoğlu and Bilge Ergün, respectively) will include patients who underwent conventional RF. In the studies, patients who underwent elective conventional radiofrequency thermocoagulation (RFT) to the articular branches of the femoral and obturator nerve were followed up for up to 6 months. The follow-up of the patients in our clinic is ongoing. In our study, the long-term follow-up of these patients will be evaluated retrospectively at 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Being over 18 years of age
2. Having received written consent
3. Those with chronic hip pain lasting longer than 3 weeks

Exclusion Criteria:

1. Major psychiatric disease
2. Patients with lumbar pressure pain or referred pain
3. Patients using anticoagulant agents
4. Patients with infection in the area to be treated
5. Those with local anesthetic allergy
6. Those with betamethasone allergy
7. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent conventional RF will be included in the prospective studies titled "Treatment of chronic hip pain with conventional radiofrequency thermocoagulation to the articular branches of the femoral and obturator nerves" and "Comparison of conventional radiofrequency thermocoagulation to the articular branches of the femoral and obturator nerves with intra-articular steroid injection and pericapsular nerve group (PENG) block in chronic hip pain" (theses of assistant Sevilay Şimşek Karaoğlu and Bilge Ergün, respectively) conducted in our clinic.
Sampling Method: Probability Sample
Enrollment: 76 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
chronic pain assessment | 12 month, 24 month
  Pain will be assessed with the SAS (Verbal Pain Score) score before surgery, at 12 and 24 months.

SECONDARY OUTCOMES:
functional capacity assesment | 12 month, 24 month
  Functional capacity will be assessed with the womac score before surgery, at 12 and 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Adnan Menderes University, Research hospital, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided